CLINICAL TRIAL: NCT00051506
Title: ALIMTA(Pemetrexed)/Cisplatin and ALIMTA(Pemetrexed)/Carboplatin in Extensive Stage Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 7210; H3E-US-JMFW; NCT00062088 (obsolete NCT alias)
Record Dates: First submitted 2003-01-10; First posted 2003-01-14 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; Carboplatin; Cisplatin

INTERVENTIONS:
Drug: ALIMTA
Drug: carboplatin
Drug: cisplatin

SUMMARY:
The purpose of this study is to evaluate the effects (good and bad) of ALIMTA plus Carboplatin or ALIMTA plus Cisplatin on you and your small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of extensive stage small cell lung cancer and can be treated with chemotherapy.
* Have received no prior chemotherapy for your disease.
* Have at least one measurable lesion.
* have an adequate performance status.
* Sign an informed consent form.

Exclusion Criteria:

* Have previously received chemotherapy for your lung cancer.
* Have been treated with a investigational drug within the last 30 days. Have previously completed or withdrawn from this study or any other study investigating ALIMTA.
* Have received radiation therapy within the last 1-2 weeks.
* Have brain metastasis that is uncontrolled.
* Have active infection or other serious condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Springdale, Arkansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Latham, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Burlington, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Charleston, South Carolina